CLINICAL TRIAL: NCT01147679
Title: Study of Social Behavior and Emotion in Frontotemporal Dementia, Alzheimer's Disease and Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mario F. Mendez, Professor of Neurology and Psychiatry, University of California, Los Angeles
Other Study IDs: 1R01AG034499 (NIH); UCLA IRB#10-001097 (Other: UCLA Institutional Research Board); R01AG034499 (NIH)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Frontotemporal Dementia; Frontotemporal Degeneration; Alzheimer's Disease; Social Behavior
Keywords: Frontotemporal dementia; Alzheimer's disease; Young-Onset; Frontotemporal degeneration; control; social; behavior; observation; emotion; morality; dementia; brain; relationships; caregiver; MRI; neurology
MeSH Terms: conditions — Frontotemporal Dementia; Alzheimer Disease; Social Behavior; Behavior; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- bvFTD: This group will include 33 patients who have been diagnosed with behavioral variant frontotemporal dementia by Dr. Mario Mendez. Patients diagnosed elsewhere must have a secondary evaluation at the UCLA FTD Clinic to confirm their diagnosis before study enrollment.
- Alzheimer's disease: This group will include 33 patients who have been diagnosed with clinically probable Alzheimer's disease by Dr. Mario Mendez. Patients diagnosed elsewhere must have a secondary evaluation at the UCLA FTD Clinic to confirm their diagnosis before study enrollment.
- Controls: 33 health individuals without clinically significant cognitive impairments will be enrolled in this study.

SUMMARY:
This study is designed to document the loss of sociomoral emotions (like empathy, guilt, and embarrassment) in patients with behavioral variant frontotemporal dementia. The loss of these emotions, which function as the motivators for social behavior, will manifest in specific interpersonal behaviors. These behaviors will correlate with regional changes in regional changes in medial frontal and anterior temporal lobes. These social and emotional changes will be compared with a young-onset Alzheimer's disease comparison group.

DETAILED DESCRIPTION:
Frontotemporal dementia (FTD) is a devastating disorder and one the most common neurodegenerative diseases in middle age. The most prominent early manifestations of bvFTD ("behavior variant" FTD) are not the memory and other cognitive deficits typical of Alzheimer's disease (AD) but, rather, disturbance in social or interpersonal behavior. A basic manifestation of this disorder is a disturbance in the emotions and motives that drive social and moral behavior. In fact, bvFTD is an incredible window to the neuroscience of social behavior. This study will help clarify the neurobiological substrates of sociomoral emotions and their associated clinical features. The findings of this proposal can have major implications for understanding the interaction between brain and social behavior and for designing future research on the basic mechanisms of social neuroscience. This research aims to document the loss of sociomoral emotions (SME) compared to primary emotions in patients with bvFTD vs. patients with AD and normal controls. We need to show that these findings are specific to bvFTD and not present in Alzheimer's disease or normal controls. The project consists of three integrated parts: 1) behavioral measures that include observations in naturalistic settings, behavioral experiments, and behavioral scales; 2) psychophysiological reactivity (i.e., measures of heart rate, blood pressure changes, galvanic skin response, facial electromyography, and facial temperature) to social and emotional stimuli; and 3) brain localization of changes in sociomoral emotions with magnetic resonance imaging technology.

ELIGIBILITY:
Inclusion Criteria (FTD or AD patients):

* The core diagnostic features of bvFTD or NINCDS-ADRDA criteria for clinically probable AD
* Mild-moderate cognitive and functional severity defined as an MMSE >/=10 and a CDR </=2.0
* Able to understand and complete procedures and to take part in the tests by hearing and understanding instructions and by seeing the stimuli to be responded to
* Willingness and ability to provide informed consent; Informed consents from caregiver and patient
* English speaking, having acquired English prior to age 13 and using it as primary language
* Minimally impaired language (language and semantics tests cut-off scores)
* Medically stable (defined as absence of medical illness that would interfere with the subject's ability to understand and participate in study procedures)
* Absence of a neurological or psychiatric illness other than bvFTD or clinically probable ADB
* Absence of cortical infarction, other cortical lesion, or significant subcortical lesion on MRI of brain
* Absence of potentially confounding medications, particularly those with effects on the peripheral nervous system, cardiovascular agents, and β-blockers
* Presence of a caregiver who can facilitate participation in this project. (see below) Where there is more than one caregiver, every effort is made to designate the closest relative as the main caregiver.

Exclusion Criteria (FTD or AD patients):

* Violation of any of the criteria above.

Inclusion Criteria (Study Partners/Caregivers):

* Personally visit and interact with the subject at least one time each week for one hour.
* Accompany the subject to each visit.
* Provide opinions about the subject's thinking (i.e., memory, language, problem-solving ability), daily activities (i.e., dressing, hygiene, mobility, household chores, and hobbies), and behavior (i.e., mood, sleep patterns, appetite, participation in social interactions).
* Share personal information including feelings of distress about the subject's behavior or feelings of burden by caregiving responsibilities.
* Read, understand and speak English fluently in order to ensure comprehension of informed consent form and informant-based assessments of the subject.
* Provide full written informed consent on his/her own behalf prior to the performance of any protocol-specific procedure.
* In the opinion of the investigator, the study partner will be compliant with the protocol and have a high probability of completing the study

Exclusion Criteria (Study Partners):

* Violation of any of the criteria above.

Inclusion Criteria (Control Participants):

* Denies neurological or psychiatric illness.
* Not currently a caregiver for a dementia patient (for at least one year).
* Does not take potentially confounding medications, including most of those with effects on the central nervous system and peripheral nervous system, cardiovascular agents, and β-blockers. The use of these medications will be assessed during a telephone screening.

Exclusion Criteria (Control Participants):

* Violation of any of the criteria above.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients evaluated by Dr. Mario Mendez at the UCLA Frontotemporal Dementia Clinic
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-09 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Psychophysiological Reactivity | within three months of study enrollment
  We will evaluate autonomic (sympathetic and parasympathetic) nervous system reactivity to sociomoral vs. non-social stimuli using measures of heart rate (and heart rate variability), blood pressure (and baroreflex sensitivity), finger pulse volume, and skin conductance changes. Investigators present social and non-social pictures, videos, and written scenarios to all three groups while recording these psychophysiologic measures.
Behavioral Reports and Observations | within three months of study enrollment
  This proposal will use methods of ethnography to classify the social behavior of bvFTD and AD patients and their caregivers in their homes and during research visits. Four social behavioral experiments or vignettes will be used to cross-validate the results of augmented participant observation. Behavioral scales will record differences between caregiver and patient assessments of behavior and further validate the results of the participant observation.
MRI Brain-Mapping | within three months of study enrollment
  An MRI scan evaluated with state-of-the-art techniques will yield three dimensional maps of localized structural changes that reflect the regions involved in mediating social, moral, and emotional behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Mendez, MD, PhD, Principal Investigator — University of California, Los Angeles; Veteran's Health Administration, West Los Angeles
Locations (1):
- UCLA Department of Neurology, Los Angeles, California, United States

REFERENCES:
- See also: The website of the Association for Frontotemporal Degeneration — http://www.theaftd.org